CLINICAL TRIAL: NCT04888897
Title: A Mixed Methods Study Investigating the Experiences, and Information and Support Needs, of People Prescribed Opioids, and the Role of Community Pharmacy
Brief Title: The Experiences of People Prescribed Opioid Pain Medicines
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Boots UK (Unknown); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21009; 289857 (Other: IRAS)
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Pain; Opioid Use
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Opioids are morphine-type medicines which come from the opium poppy or are similar-to morphine. They are very effective for short-term pain, cancer pain, and pain at the end of life. Opioids are thought to be less useful for treating long-term non-cancer pain. Side effects are common and can be serious. People who take opioids for longer periods are at risk of tolerance (needing a higher dose to get the same effect), dependence (unable to cut down or stop without withdrawal effects), and addiction (uncontrollable use despite harmful consequences).

In the UK, opioid prescribing has increased substantially over the last two decades. Doses are higher and opioids are taken for longer, suggesting many people are at risk of harmful effects without useful pain relief. Research into opioid dependence and addiction has found people do not always fully understand the risks of these medicines at the start of treatment. Local Community Pharmacists could be used to improve information and support for those prescribed opioids.

This study aims to get a better understanding of the experiences of people prescribed opioids and their information and support needs, and to investigate whether information and support could be improved using Community Pharmacists. Findings may improve care for people prescribed opioids in the future.

The study will involve questionnaires and interviews with adults prescribed an opioid medicine for pain, not caused by cancer, over a period of at least 3 months. Participants will be recruited from GP practices in England.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Adults aged 18 years and above, with no upper age limit
* Prescribed any opioid analgesic (defined as any opioid or opioid/paracetamol combination analgesic from sections 4.7.2 and 4.7.1 British National Formulary) for non-cancer pain for a period of ≥3 months (defined as ≥ 2 opioid prescriptions issued in the previous 3 months with a minimum interval of 60 days between the first and last prescription)

Exclusion Criteria:

* Cancer pain
* Terminal illness
* Vulnerable patients (e.g. severe mental illness, learning difficulties, dementia, care home residents)
* Unable to understand English
* Deemed by their GP to be inappropriate to contact

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients registered with a GP practice in England who have been prescribed an opioid medicine for non-cancer pain by their GP over a period of at least 3 months. Purposive sampling of GP practices within the NIHR CRN East Midlands is planned. We aim to utilise a sample of practices with a range of characteristics which are representative of GP practices across the East Midlands.
Sampling Method: Non-Probability Sample
Enrollment: 619 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
To identify whether people prescribed opioids for non-cancer pain need more information and support at the start of treatment. | 6 -12 months
  The information and support needs of patients will be explored through the study questionnaire and interviews.

SECONDARY OUTCOMES:
To assess and explore the difficulties experienced by people prescribed opioids for non-cancer pain. | 6 - 12 months
  Determined by the Prescribed Opioid Difficulties Scale (PODS) within the study questionnaire and qualitative interviews.
To explore the perceptions of people prescribed opioids for non-cancer pain on the information they received and the need for improved information and support at the start of treatment | 6 -12 months
  Explored through related items in the questionnaire and qualitative interviews.
To investigate the use of pharmacy by people prescribed opioids for non-cancer pain and their views on using community pharmacists to provide additional information and support for opioid pain medicines | 6 -12 months
  Explored through related items in the questionnaire and qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Boyd, PhD, Principal Investigator — Associate Professor, University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No